CLINICAL TRIAL: NCT00515697
Title: Phase II Single Arm Study of IMC-1121B in Patients With Metastatic Renal Cell Carcinoma With Disease Progression on or Intolerance to Tyrosine Kinase Inhibitor Therapy
Brief Title: A Study of Ramucirumab in Participants With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13921; I4T-IE-JVBP (Other: Eli Lilly and Company); CP12-0605 (Other: ImClone Systems)
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab (Experimental): Intravenous infusion at 8 milligrams per kilogram (mg/kg) on day 1 of every 14-day cycle.
  Interventions: Biological: Ramucirumab

INTERVENTIONS:
Biological: Ramucirumab — Ramucirumab is an injectable solution administered as an intravenous infusion over 1 hour at a dose of 8 mg/kg day 1 of every 14-day cycle.
  Other Names: IMC-1121B; LY3009806

SUMMARY:
The purpose of this study is to determine whether ramucirumab is effective treatment in participants with metastatic renal cell carcinoma who have developed progressive disease or become intolerant to tyrosine kinase inhibitor therapy.

DETAILED DESCRIPTION:
The Primary objective is to determine the best objective response rate (ORR) of ramucirumab when administered to participants with metastatic renal cell carcinoma (RCC) whose disease has progressed during therapy with a tyrosine kinase inhibitor (TKI, sunitinib and/or sorafenib) or who have developed intolerance to these agents.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed clear cell RCC
* The participant is ≥ 18 years of age
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1 or Karnofsky Performance Status (KPS) ≥ 80%
* The participant has had a prior nephrectomy (as therapy for RCC)
* The participant has metastatic RCC
* The participant has a life expectancy of > 3 months
* The participant has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* The participant has received prior therapy with a TKI (sunitinib and/or sorafenib) with either disease progression on TKI therapy (progression within 60 days of the last dose of TKI) or intolerance to TKI (unable to continue therapy because of side-effects). A participant with progression during a protracted treatment break is not eligible unless the participant has had progression or intolerance as defined above
* The participant has resolution of all clinically significant toxic effects of prior cancer therapy to grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0 (NCI-CTCAE)
* The participant has adequate hematological functions [absolute neutrophil count (ANC) ≥ 1500 cells per milliliter (cells/mL), hemoglobin ≥ 9 grams per deciliter (g/dL) and platelets ≥ 100,000 cells/mL]
* The participant has adequate hepatic function [bilirubin within normal limits (WNL), aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN), or ≤ 5.0 times the ULN if the transaminase elevation is due to liver metastases]
* The participant has normal renal function or mild renal dysfunction [creatinine ≤ 2.2 milligrams per deciliter (mg/dL)]
* The participant's urinary protein ≤ 1+ on dipstick or routine urinalysis [(UA); if urine dipstick or routine analysis is ≥ 2+, a 24-hour urine for protein must demonstrate < 1000 (milligrams) mg of protein in 24 hours to allow participation in the study]
* The participant must have adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.8 and a partial thromboplastin time (PTT) ≤ 1.5 X ULN. Participants on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight (LMW) heparin and if on warfarin must have a INR between 2 and 3 and have no active bleeding or pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or known varices)
* The participant is able to provide informed written consent
* The participant , if sexually active, is postmenopausal (last menstrual period > 2 years prior to study), surgically sterile, or is using effective method of contraception in the opinion of the investigator
* The participant , if female, must have a negative serum pregnancy test upon entry into this study
* The participant has a normal thyroid stimulating hormone (TSH) value. Participants with an abnormal TSH may be eligible provided they meet all other eligibility criteria and have ECOG performance status 0-1. Participants with an abnormal TSH value require a full thyroid evaluation prior to enrollment. Endocrinology consultation may be performed at the discretion of the investigator
* The participant has serum calcium within normal limits

Exclusion Criteria:

* The participant has received prior treatment with bevacizumab
* The participant has known brain or leptomeningeal metastases
* The participant has received >2 prior cytotoxic chemotherapy regimens for RCC
* The participant has received antitumor therapy (biologic agents, major surgery, or investigational agent) within 28 days prior to enrollment on study. The participant has received radiation therapy within 14 days prior to enrollment on study. Participants with metastasis in weight bearing bones at high risk for pathologic fracture may participate provided that appropriate surgical intervention and/or radiation therapy is undertaken and completed at least 28 days prior to enrollment
* The participant has received > 1 prior bio-immunotherapy regimens (defined as either interleukin-2 or interferon alpha given as monotherapy, concurrently, or sequentially as planned)
* The participant has a concurrent active malignancy other than adequately treated non-melanomatous skin cancer or other non-invasive carcinoma or in situ neoplasm. A participant with previous history of malignancy is eligible, provided that he/she has been disease free for > 3 years
* The participant has a nonhealing wound or ulcer
* The participant has a known alcohol or drug dependency
* The participant is pregnant or breastfeeding
* The participant has a coexisting medical or psychiatric problem of sufficient severity to limit compliance with the study and/or increase the risks associated with study participation or study drug administration or interfere with the interpretation of study results
* The participant has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders in the opinion of the investigator
* The participant has known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (11):
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Flemington, New Jersey
  - ImClone Investigational Site, Buffalo, New York
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Drexel Hill, Pennsylvania
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Arlington, Texas
  - ImClone Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study comprised 3 study periods: pretreatment, treatment, and (posttreatment) follow-up. 40 participants signed the informed consent.
Groups:
- Ramucirumab: Ramucirumab at 8 milligrams per kilogram (mg/kg) infused intravenously over 1 hour, on Day 1 of every 14-day cycle. Treatment continued until there was evidence of disease progression or intolerable toxicity.
Period: Overall Study
Arm/Group | Ramucirumab
Started | 39
Received at Least 1 Dose of Study Drug | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: participants who received any quantity of ramucirumab.
Arm/Group | Ramucirumab
Number analyzed (Participants) | 39
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 27
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 35
  Black or African American | 3
  Asian | 1
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  More than one race | 0
Region of Enrollment [Number; unit: participants]
  United States | 39
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (Objective Response Rate)
Description: The percentage of participants with a best overall response of confirmed complete response (CR) or partial response (PR) as classified according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. CR is the disappearance of all target and non-target lesions and normalization of tumor marker levels. PR is having at least a 30% decrease in the sum of the longest diameter of target lesions without new lesions and progression of non-target lesions. The percentage of participants with objective response=(number of participants whose best overall response during therapy is CR or PR/number of participants treated)*100.
Time Frame: First dose to date of objective progressive disease or death due to any cause (up to 34 months)
Population: Intent-to-treat population: participants who received any quantity of ramucirumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 39
percentage of participants | 5.1 [0.6 to 17.3]

2. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is measured from the date of the first dose to the first documented date of disease progression as classified according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria or death from any cause. Disease progression is having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of a new lesion. Data for participants whose disease does not progress or for whom no post-baseline assessment is made are censored at the day of their last tumor assessment. Data for participants whose disease does not progress who are subsequently lost to follow-up are also censored at the day of their last tumor assessment.
Time Frame: First dose to measured progressive disease or death due to any cause (up to 34 months)
Population: Intent-to-treat population: participants who received any quantity of ramucirumab. The number of participants censored was 4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab
Number analyzed (Participants) | 39
months | 7.1 [4.1 to 9.7]

3. Secondary Outcome: Percentage of Participants Showing Disease Control at Week 12
Description: Participants who were alive and did not experience disease progression were considered to have disease control at 12 weeks. Disease control was based on lack of disease progression using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. According to RECIST criteria, disease progression was having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of non-target lesion and/or detection of new lesion. Participants whose disease progression was symptomatic were not considered to have disease control. The percentage of participants showing disease control=(number of participants who did not have disease or symptomatic progression at Week 12/number of participants treated)*100.
Time Frame: Week 12 [Cycle 6 (1 cycle=14 days)]
Population: Intent-to-treat population: participants who received any quantity of ramucirumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 39
percentage of participants | 64.1 [47.2 to 78.8]

4. Secondary Outcome: Percentage of Participants With Objective Response (Objective Response Rate) at 12 Weeks
Description: The percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) at Week 12, as classified according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. CR is the disappearance of all target and non-target lesions and the normalization of tumor marker levels. PR is having at least a 30% decrease in the sum of the longest diameter of target lesions without new lesions and progression of non-target lesions. The percentage of participants with objective response=(number of participants whose best overall response achieved at 12 weeks was CR or PR/number of participants treated)*100.
Time Frame: Week 12 [Cycle 6 (1 cycle=14 days)]
Population: Intent-to-treat population: participants who received any quantity of ramucirumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 39
percentage of participants | 0.0 [0.0 to 9.0]

5. Secondary Outcome: Median Duration of Overall Response
Description: Duration of response is the interval from the date of initial documented response [confirmed complete response (CR) or partial response (PR)] to the first documented date of disease progression as classified according to Response Evaluation Criteria In Solid Tumors (RECIST version 1.0) criteria, or initiation of other (or additional) antitumor therapy is first reported, or death due to any cause. CR is the disappearance of all target and non-target lesions and the normalization of tumor marker levels. PR is having at least a 30% decrease in the sum of the longest diameter of target lesions without new lesions and progression of non-target lesions. Disease progression is having at least a 20% increase in the sum of the longest diameter of target lesions and/or unequivocal progression of a non-target lesion and/or detection of a new lesion. Data from participants who did not relapse were censored on the day of their last tumor assessment.
Time Frame: Time of first response (CR or PR) to disease progression, initiation of other (or additional) antitumor therapy, or death due to any cause (up to 34 months)
Population: Participants who received any quantity of ramucirumab and had confirmed complete response or partial response. The number of participants censored was 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab
Number analyzed (Participants) | 2
months | NA [2.8 to NA] — Two participants had confirmed response (1 CR and 1 PR, both occurring more than 12 weeks after starting drug therapy). The participant with CR did not relapse and data were thus censored for the analysis.

6. Secondary Outcome: Minimum Concentration (Cmin) of Ramucirumab
Time Frame: Immediately prior to the Week 32 infusion treatment [Cycle 16 (1 cycle=14 days)]
Population: Participants who received any quantity of ramucirumab and had evaluable pharmacokinetic data at the specified time point.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Ramucirumab
Number analyzed (Participants) | 11
micrograms per milliliter (mcg/mL) | 147 (76.2)

7. Secondary Outcome: Maximum Concentration (Cmax) of Ramucirumab
Time Frame: 1 hour after the end of the Week 32 infusion treatment [Cycle 16 (1 cycle=14 days)]
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Ramucirumab
Number analyzed (Participants) | 9
micrograms per milliliter (mcg/mL) | 595 (239)

8. Secondary Outcome: Summary Listing of Participants Reporting Drug-Related Treatment-Emergent Adverse Events
Description: Data presented are the number of participants who experienced treatment-emergent adverse events (TEAE), serious adverse events (SAE), Grade 3 or 4 TEAE, or adverse events (AE) leading to discontinuation of treatment that were considered to be related to ramucirumab. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: First dose to study completion (up to 34 months) plus 30-day safety follow-up
Population: Intent-to-treat population: participants who received any quantity of ramucirumab.
Measure: Number; unit: participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 39
participants
  Related TEAE | 37
  Related SAE | 6
  Related Grade 3 or 4 TEAE | 10
  Related AE leading to discontinuation | 7

ADVERSE EVENTS:
Arm/Group | Ramucirumab
Serious Adverse Events (participants affected / at risk) | 12/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=39)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) — This event resulted in death.
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 (8)
VISION BLURRED (Eye disorders) | 2 (2)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 (3)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (9)
CONSTIPATION (Gastrointestinal disorders) | 8 (9)
DIARRHOEA (Gastrointestinal disorders) | 7 (16)
DYSPEPSIA (Gastrointestinal disorders) | 2 (3)
ERUCTATION (Gastrointestinal disorders) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 10 (13)
TOOTHACHE (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 9 (10)
CHILLS (General disorders) | 6 (7)
FACE OEDEMA (General disorders) | 2 (2)
FATIGUE (General disorders) | 19 (37)
INFUSION RELATED REACTION (General disorders) | 3 (6)
OEDEMA PERIPHERAL (General disorders) | 14 (19)
PYREXIA (General disorders) | 2 (2)
PHARYNGITIS (Infections and infestations) | 3 (7)
RHINITIS (Infections and infestations) | 7 (14)
SINUSITIS (Infections and infestations) | 2 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5)
CONTUSION (Injury, poisoning and procedural complications) | 3 (3)
BLOOD CREATININE INCREASED (Investigations) | 4 (5)
WEIGHT DECREASED (Investigations) | 6 (8)
WEIGHT INCREASED (Investigations) | 3 (3)
ANOREXIA (Metabolism and nutrition disorders) | 10 (13)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 (5)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (16)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (11)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5)
DIZZINESS (Nervous system disorders) | 4 (6)
HEADACHE (Nervous system disorders) | 14 (38)
NEUROPATHY (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 (3)
SOMNOLENCE (Nervous system disorders) | 2 (2)
ANXIETY (Psychiatric disorders) | 4 (4)
DEPRESSION (Psychiatric disorders) | 2 (3)
INSOMNIA (Psychiatric disorders) | 4 (4)
HAEMATURIA (Renal and urinary disorders) | 2 (2)
PROTEINURIA (Renal and urinary disorders) | 7 (10)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (13)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (11)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 13 (19)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (5)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (5)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2 (2)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 (4)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (11)
RASH (Skin and subcutaneous tissue disorders) | 4 (5)
HYPERTENSION (Vascular disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.